CLINICAL TRIAL: NCT06533293
Title: Promoting Functional Neck Motion in Patients With Cerebral Palsy Using a Dynamic Neck Brace
Brief Title: Improving Neck Control in Children With Cerebral Palsy Using Robotics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: New York Medical College (Other)
Responsible Party: Principal Investigator, Sunil Agrawal, Professor, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAV1209
Record Dates: First submitted 2024-06-08; First posted 2024-08-01 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Palsy; Neck Disorder
Keywords: Motor training, Robotics
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Masking Description: This is an exploratory study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Device (Experimental): Motor learning principles will be combined with robotics to apply gentle forces on the head-neck during training.
  Interventions: Device: Neck Brace Device

INTERVENTIONS:
Device: Neck Brace Device — The neck brace device will be manufactured in the Mechanical Department at Columbia University. The device measures head motion and EMG by electronic sensors, passively supports the head in certain configurations by springs, and actively assists head movement by motors.
  Motor learning principles will be combined with robotics to apply gentle forces on the head-neck during training.

SUMMARY:
The goal of this study is to characterize the head-neck motion of children with cerebral palsy and investigate how robotics can be used to improve the head-neck coordination of these children.

Aim 1 is a cross-sectional study. In this single-session, kinematic and muscle activity data will be collected during the postural static, active-proactive, and reactive postural head tasks. Gross Motor Functional Classification System (GMFCS) levels will also be collected to categorize the sample into subgroups.

Aim 2 is a prospective cohort quasi-experimental study. The data will be collected at baseline, across 12 intervention sessions, 1 week post-intervention, and 3 months follow-up.

Functional assessments will be used to compare across the pre, mid, and post training. Participants will be assessed in Gross Motor Functional Measures (GMFM), Seated Posture and Reaching Control (SP&R-co), and Canadian Occupational and Performance Measure (COPM). The primary outcomes will be SP&R-co test and COPM pre- and post-intervention.

DETAILED DESCRIPTION:
The study investigators plan to recruit a sample of 30 children and adults (10 able-bodied children/young adults for the characterization phase and 20 children/young adults with bilateral cerebral palsy: 10 classified as GMFCS IV and 10 classified as GMFCS V). These participants will be aged 11-21 years.

A motion capture/body mounted sensors and Electromyography (EMG) system will be used for measurement. This study will utilize specialized robotics that can apply gentle forces on the head-neck during movement training using the principles of motor learning.

ELIGIBILITY:
Inclusion Criteria:

* CP, as medical diagnosis
* GMFCS IV-V classification

Exclusion Criteria:

* severe cognitive deficits
* uncontrolled epilepsy
* severe dyskinesia
* spinal cord malformations
* severe vertebral column deformities (scoliosis >40° and/or kyphosis >45º)
* blindness
* chemo-denervation 3 months before study

Ages: 11 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Seated Postural and Reaching Control (SP&R-co) | Data will be collected at baseline, immediately after post-intervention, 1 week post-intervention, and 3 months follow-up.
  Measurement of head-trunk and reaching control of children and young adults with CP while sitting static, active, proactive, and reactive postural dimensions while providing support at different regions of the torso.

SECONDARY OUTCOMES:
Gross Motor Functional Measure-items set (GMFM-IS) | Data will be collected at baseline, immediately after post-intervention, 1 week post-intervention, and 3 months follow-up.
  This is an abbreviated version of the original GMFM-66 to measure the gross motor status of the children with CP across 5 dimensions: A) lying and rolling, B) Sitting, C) Crawling and Kneeling, D) Standing and E) Walking, Running and Jumping.
Canadian Occupational Performance Outcome (COPM) | Data will be collected at baseline, immediately after post-intervention, 1 week post-intervention, and 3 months follow-up.
  Measurement of perceived parent- and child-based goals and preferences that are specific to motor impediments that restrict participation.

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Agrawal, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - ROAR Lab, Mudd Hall, New York, New York
  - Columbia University Irving Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No
This is a exploratory study at this point.

REFERENCES:
- See also: Amyotrophic lateral sclerosis patients regain head-neck control using a powered neck exoskeleton — https://scholar.google.com/citations?view_op=view_citation&hl=en&user=zavGyr4AAAAJ&cstart=20&pagesize=80&sortby=pubdate&citation_for_view=zavGyr4AAAAJ:j7XjBeKFbTsC